CLINICAL TRIAL: NCT02592304
Title: Preoperative Assessment of Mesorectal Lymph Nodes by Dual Energy CT. PUMK-DECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Issam al-Najami, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SvG2-4-13-07
Record Dates: First submitted 2015-10-07; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dual energy ct (Other)
  Interventions: Device: Dual energy computed tomography

INTERVENTIONS:
Device: Dual energy computed tomography — one extra scanning with a dual energy ct.

SUMMARY:
Endpoints subproject 1: To develop a reproducible method for the detection of lymph nodes by DECT in operation specimens from rectal resection for cancer. sub project 2: Primary endpoint: To evaluate the sensitivity and specificity for malignant lymph nodes in vitro RC specimens compared with histopathology. Secondary endpoint: To assess DECT as imaging tool for the diagnosis of malignant lymph nodes at RC. Histopathology will be used as reference.Subproject 3: Primary endpoint: To compare the sensitivity, specificity, positive- and negative predictive values, accuracy of DECT and standard MRI. Secondary: To evaluate the value of the gold standard for the use of imaging methods for the description of the lymph node, validated by histopathology. Secondary: to determine the value of tumor diagnostics using DECT.subproject 4: To assess the value of DECT as imaging tool for diagnosing response to chemo radiotherapy of malignant lymph nodes.

DETAILED DESCRIPTION:
Background Long-term survival for patients with cancer of the rectum (RC) is through the last 20 years dramatically improved from about 30% to 65% . Overall focus on disease with the creation of multidisciplinary teams, national quality databases certification of surgeons, etc. have contributed to the development especially in the last 10-15 years . The introduction of pre-operative Oncology, known as neoadjuvant treatment increased the survival rate by up to 10% in certain patient series. However, the prognosis remains poor for advanced cases, qua risk of metastasis and local cancer relapse.

Surgical treatment remains the cornerstone of curative treatment of RC. Total mesorectal excision (TME) includes resection of both the tumor and the surrounding mesorectal fat. TME is currently used as the gold standard for surgical treatment of RC. The use of TME has reduced local relapse rate to less than 10%.

TME surgery combined with preoperative chemotherapy and radiation therapy if the cancer is in an advanced stage (T3), and often with high-dose radiotherapy and chemotherapy in the most advanced cases of T-stage 4.

Complications of TME are present in more than 40% of patients. Most often in the form of wound dehiscence, infection, sexual dysfunction, bowel disorders and the necessity of a stoma. More than 50% of patients have permanently reduced quality of life.

Minimally invasive therapies (trans-anal endoscopic microsurgery (TEM)) for the curative treatment of early rectal cancers, is well-validated. The complication rate is low, and above all, the operative mortality of less than 1% even in the elderly and patients with comorbidities, opposed to 10% at standard surgery. The use of TEM surgery early in the rectum cancers in selected patients will thus be able to reduce the risk of complications and improve the overall long-term survival. Even though the disease-specific survival is reduced due to a less radical procedure. The Danish screening program for colorectal cancer will result in a significant increase in the detection of early cancers.

Thus, over the past 10-15 years, there is developed a complex treatment algorithm with tailored surgery, in combination with oncological treatment if necessary. The full benefits of the available treatment options require that you pre-treatment, stage classify the disease so the patient can be allocated to the proper treatment. The tumor extent of ingrowth into the different layers in the rectum (T-stage) can now be carried out with great certainty preoperatively.

Patients with tumor stage T1 may be candidates for TEM surgery because only 10% of these patients have metastases to the lymph nodes. Cancers of the stage T2 may be candidates for TEM if they have increased operative mortality risk. A local resection of the cancer is of course undesirable, in the lymph node metastases as they are not included in the resection. Distant metastases can with certainty be detected with CT and MRI scans. Preoperative assessment of lymph node involvement is difficult and uncertain for daring to use it to allocate candidates for local resection.

The indication for TEM treatment of rectal cancers can potentially be extended if you could allocate patients independent of tumor stage - based on lymph node stage.

The detection of disease spread to the lymph nodes has a decisive impact on the choice of treatment modality. Moreover the impact on prognosis and local recurrence.

1. Local resection performed only for N0.
2. The number of involved lymph nodes has a prognostic value for the outcome of surgery for RC.
3. Detection of tumor cells in the lymph nodes at the mesorectal fascia (which forms circumferential resection margin CRM) increases the risk of recurrence. Patients must have neoadjuvant oncological treatment.
4. Lymph nodes located outside the mesorectal fascia may require extended lymphadenectomy, to achieve a good oncological outcome and avoid relapse.

Today, magnetic resonance scan (MRI) and trans rectal ultrasound (TRUS) is used as the gold standard in the imaging staging of RC. Studies have demonstrated high specificity for the assessment of T stage and CRM using the preoperative MRI. Comparative high specificity is obtained in the intermediate hands with TRUS.

In contrast to T stage and CRM classification, the MR and TRUS have shown poor results compared to N-staging of RC. Even worse results arise for the use of conventional Computed Tomography Scan (CT) for lymph node diagnostics, with a median sensitivity of 80% (from 62.5 to 91.9%) and median specificity of 77.8% (50- 87.9%).

Research should be directed towards improvement of lymph node diagnostics by RC, in order to take full advantage of the differentiated treatments.

Dual Energy Computed Tomography (DECT) is an imaging modality, which in recent years has gained a foothold in the diagnosis of several types of micro-lesions. DECT provides information on a tissue reaction when it is affected by different energy levels. This gives you information about its composition, based on the known K-edge value of different substances. K-edge is defined by the maximum visual attenuation of a substance in a DECT scan when it is affected by a certain amount of energy. The energy required to achieve a given k-edge depends on the individual substances atomic size, and therefore increases with the atomic mass.

The technique is known from, for example, kidney stones diagnosis, pancreatic cancer staging, vascular anomalies such as classification of aortic aneurysms, detection of coronary plaques etc.

A study from 2013 by Zalai Pan et al investigated the association between histologically confirmed gastric cancer, and the discovery of metastatic lymph nodes by DECT. Ninety-six patients were included. Two groups of radiologists were blinded to the endoscopic and histological findings. Lymph nodes of 6 mm were included in the N-staging. They found a sensitivity of 85.4% for N0, 84.4% N1, 91.7% N2. Furthermore, it showed a significant difference in the uptake of iodine (from the iodine-containing contrast) with the K-edge value of 33.20 keV, in malignant and non-malignant lymph nodes.

Thus, there is the hope of both iodine and Gadolinium found in X-ray contrast agent, is absorbed in cancer tissues, and gives a recognizable signal in dual energy CT scanning.

. Hypotheses

1. It is possible to develop a standardized method for DECT scanning of the rectum specimens, removed during surgery.
2. Metastatic lymph nodes suspected by DECT can be verified histopathological.
3. DECT can increase the sensitivity and specificity of the diagnosis of lymph node compared to other imaging modalities.
4. The effect of chemo-radiotherapy to the lymph nodes can be detected by DECT

Study Design The study is a prospective observational study, based on patients with newly diagnosed rectum cancer at the Surgical Department A, Odense University Hospital.

Patients will automatically be divided into 3 groups according to the preoperative stratification, in a group which will refer to the direct operation either TEM (group 1) or TME (GROUP2) after the preoperative imaging staging, and a group of 3 which will undergo two imaging phases, before and after the radio or chemo-radiotherapy before surgery.

Methods Subproject 1: In Vitro DECT scan of rectal specimens. Subproject 1 scan without contrast

Part 1 procedure: 3 patients with visible lymph nodes in the perirectal fat tissue by MRI are selected.

Scenario 1 - after TME the specimens will be transported to the pathological institute for the preparation of 3mm. thick sections from the distal to the proximal resection rim.

* The product is placed in an aluminum lattice.
* All cuts of 3 mm gets numbered and photographed.
* The ex-vivo specimen scan is done; this is done in three different ways to determine the ideal technique.

  1. specimen is scanned between 2 gel plates
  2. specimens is scanned in the air
  3. specimens is scanned in flooded container
* All sections of 3 mm which is photographed and numbered, gets coupled with its DECT-scan image.
* The specimens are placed in formalin, and the same scans will be made 24 hours later. This is to compare the effect of formalin on the DECT scans of specimens.
* The ideal technique for the in vitro DECT scan of specimens will be determined.

The scan with contrast

Second part procedure: Nine patients with visible lymph nodes in the perirectal fat tissue by MRI will be selected.

* At the preparing meeting with the patients in KA (surgical day center, Svendborg), the patients will receive information about the study, provided written material, and consent will be obtained.
* questions in time from the information in KA, to participation in the study to time of surgery, may be directed to the investigator. The investigator is present at the time of surgery, and can take questions from the patient.
* Upon written consent from the patients the following procedure will be completed:

  1. 5 min. before the default central ligating of a. mesenteric inf. three patients will receive iv, iodine-containing contrast media, Omnipaque 350 mg iodine / ml, a total of 10 ml.

For 3pt: intra venous Gadovist (Gadobutrol) 1.0 mmol / ml total 0.1 mmol / kg For 3pt: using rectoscope and a needle 5 ml of 1 mmol / ml Gadovist will be administered, for examination of the sentinel node.

2. After TME the specimens are prepared and DECT scanned according to the ideal technique found by part-1 procedure.

3. All lymph nodes, designated normal or pathological by DECT scan will be analyzed by a pathologist, who is blinded to the scan results. The lymph nodes will be assessed under the gold standard for pathological assessment of these (38). In this process it is possible to remove the lymph node for histopathological validation, as they are numbered according to photograph and scan images.

4. Pathologist fills in Annex 2 5. Investigator assesses DECT scan pictures, together with the radiologist. 6. Investigator fills in Annex 1

Subproject 2: assess the sensitivity and specificity of benign / malignant differentiation in DECT scanning of in Vitro rectal specimens.

* All included patients under the standardized preoperative imaging staging, by written consent, will get an additional DECT scan of the pelvis, either with Gadovist 1.0 mmol / ml, 0.1 mg / kg iv, or after administration of standard CT contrast Omnipaque. DECT scans can be performed in the same scanner and at the same session as the conventional CT of the thorax and abdomen. Images should result in ongoing 3mm thick sections of the pelvis, perpendicular to the rectum wall, from the anorectal transition to promontory level.
* Conventional CT scan of the thorax and abdomen, and MRI of the rectum will be used as usual, for the stratification of patients to appropriate treatment cf. Figure 1
* Endoscopist informs about the study and provides written material for signature when the detection of a rectal cancer is made.
* Questions from patients about participation in the study during the period between endoscopy and scanning can be directed to the investigator. The investigator is present at the time of the planned preoperative imaging staging, and accept any questions from the patient.
* Written acceptance delivered to the investigator in the preoperative imaging staging. A Copy of the acceptance will be provided the radiologist.
* Item 2-6 from subproject 1 second procedural element is repeated.

Subproject 3: Best protocol during subproject 2, compared with standard MRI of malignant lymph nodes in the mesorectum in patients who have not received neoadjuvant therapy.

* As mentioned above, the aim is the inclusion of a total of 100 pts. With RC. After the 1-year inclusion period analyzed the scanning images. All the preoperative in vivo images is reviewed by dedicated radiologists, with a particular focus on lymph node detection. Morphological criterions as used in MRI is used to determine whether a lymph node is malignant or not (39), both in the preoperative MR and DECT scanning.
* Radiologists are blinded to the results of the preoperative MRI staging and the histopathological results.
* Only patients who did not receive neoadjuvant therapy will be included in the subproject 3, radiologist fills in Annex 1.
* Investigator compares in vivo scan results.
* Investigator compares in vivo scanning results with in vitro scan results and pathology results. The results are calculated as N0, N1 or N2

Subproject 4: Evaluate DECT ability to follow changes in lymph node status of malignancy after adjuvant chemo-radiotherapy.

* Patients who have received adjuvant chemo-radiotherapy will be included.
* Following the same procedure as subproject 2 the patients are scanned a second time after adjuvant chemo-radiotherapy.
* The rescans are described according to the description procedure in subproject 3.
* Annex 1 is filled in.
* Annex 1 from before and after adjuvant radio chemotherapy will be compared.

Statistics and data analysis

Prerequisites for patient collection, for in Vitro DECT scanning after the administration of Gadovist as a contrast agent:

Median figures for the diagnosis of lymph nodes on MRI in patients with RC are as follows:

* 70% of patients with RC have no visible lymph nodes.
* 15% of patients with RC have visibly benign lymph nodes.
* 15% of patients with RC have visibly malignant lymph nodes (40). 5 shows an in average 5 lymph nodes are seen per patient.

A sample size analysis showed that a number of visible nodes 150 in total were needed to achieve a sensitivity of 70% (95% CI 56% -80%). Knowing that 5 Iymph nodes are seen in average per patient would necessitate a population of 100 pts. Included. (15% of 100) x5 Iymph nodes= 75 visible benign Iymph nodes + (15% of 100) x5 Iymph nodes = 75 visible malignant lymph nodes.

Total number of Iymph nodes = 150

Ethical considerations The project must is approved by the research ethics committees in the Region of Southern Denmark and by the Data Inspectorate in Odense university hospital /Svendborg.

First contact with the patient before inclusion in the project will take place on the day when, after having endoscopic examination, found a malignant tumor in the rectum. The patient will then be informed about the project by one of the doctors of the department, in an uninterrupted interview rooms designed for the information of patients and their relatives. Written information will be disclosed.

Patients will have a minimum of 3 days of reflection before accepting participation in the project.

When the patient accepts the participation in the project it will only be medically relevant information that will be obtained in the patient's chart. This will include age, gender, pregnancy, other diseases, allergies and information on details of the patient's cancer.

DECT scan is a painless procedure that can be done in line with the preoperative scans. Disregarding the known risks of administering the contrast agent in the form of anaphylactic reactions, patients are not exposed to medical risk. Using gadolinum based contrast agents are suspected to be contributing to nephrogenic systemic fibrosis (NSF), but there is no case of this by the recent report of Committee for Medicinal Products for Human Use (CHMP) in 2007. Allergic reactions to iodinated contrast agents are described with a frequency of 0.2%, most commonly in the form of hives. Serious adverse reactions, as anaphylactic shock is described with a frequency of 0.01%.

Patients in sub-project 1 are under the administration of contrast agent preoperatively under close surveillance by the anesthesiologists, and any possible allergic reaction could be treated immediately.

Included patients will be exposed to increased radiological radiation, equivalent to 1-10 mSv and therefore only one additional CT scan of the abdomen.

The selected specimens will be treated in exactly the same way as it is legally described in that matter. The investigator will, in the usual pathological preparation of the specimens, photograph the specimens and categorize them in the project gradient time. After completing the project, the picture material will be made anonymous.

It should be emphasized that the results of the experiments related to the scans will not to have a therapeutic impact.

Perspective In the event that the study shows that DECT enhances the quality of the imaging staging of patients with RC, the consequences will be substantial. If the accuracy of lymph node positive for RC reaches 90%, a local resection would be possible for the 10% of the lymph nodes positive T1 tumors. Furthermore you may be able to offer local resection for the 75% of T2 and T3 early cancers that have not spread, and who otherwise meet the criterions for local resection. With secure node diagnostics, the surgical oncological treatment will improve in terms of prognosis and the rate of local relapse. Furthermore, one with better lymph node diagnostics one can avoid unnecessary neoadjuvant chemo-radiotherapy to the previous false-positive patients. They are between 25 and 50%.

Medical oncology one will be able to assess the effect of chemotherapy on RC patients, with the possibility of optimizing the oncological treatment.

Opportunities for practical implementation: We have access to dual-CT and contrast. The feasibility study is completed.

Study design problems:

There is a risk of categorizing some of the lymph nodes seen on the preoperative DECT scan as false positive, if they are not found in the in-vitro scans, due to the effect of radiation therapy. However this is a fact for both MRI and DECT.

ELIGIBILITY:
Inclusion Criteria:

- All patients with an endoscopic suspected rectal cancer.

Exclusion Criteria:

* Chronic kidney failure
* pregnancy
* rectal cancer recurrence
* known contrast allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the detection of lymph nodes by DECT in specimens from rectal resection for cancer. | 6 months
  Measurments will be done in Hounsfield units, effective z-value and iodine, water and gadolinium concentrations.
sensitivity and specificity for the detection of malignant lymph nodes in vitro RC specimens compared with histopathology | 6 months
  Measurments will be done in Hounsfield units, effective z-value and iodine, water and gadolinium concentrations.
sensitivity, specificity, positive- ognegative predictive values, accuracy of DECT and standard MRI. | 1 year
  Measurments will be done in Hounsfield units, effective z-value and iodine, water and gadolinium concentrations. Histopathological proved malignant lymph nodes will be compared to histopathological proved benign lymph nodes.
DECT as imaging tool for diagnosing response to chemo radiotherapy of malignant lymph nodes, and tumors. | 1 year
  Rectal Cancer Regression Grade (RCRG) according to the three levels RCRG 1-3. RCRG 1: the tumour is either sterilised or only microscopic foci of adenocarcinoma remain; RCRG 2: marked fibrosis, but with macroscopic tumour still present; and RCRG 3: little or no fibrosis in the presence of abundant macroscopic tumour , based on measurments of Hounsfield units, effective z-value and iodine, water and gadolinium concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Issam al-Najami, Svendborg, Southern Denmark, Denmark